CLINICAL TRIAL: NCT00730054
Title: Clonidine-Remifentanil. Effect of the Combination on Acute Pain and Respiration in Healthy Volunteers
Acronym: Remiclon
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Dr. Jon Bragi Bergmann, Dep.of anasthesiology, Rikshospitalet, Oslo, Norway
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: S-03025
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-08

CONDITIONS: Acute Pain; Respiration; Sedation
Keywords: Remifentanil; clonidine; acute pain; respiration; sedation; cognitive function
MeSH Terms: conditions — Acute Pain; Respiratory Aspiration | interventions — Remifentanil; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Clonidine
  Interventions: Drug: Remifentanil+clonidine
- 2 (Active Comparator): Remifentanil
  Interventions: Drug: Remifentanil+clonidine
- 4 (Experimental): Remifentanil+clonidine
  Interventions: Drug: Remifentanil+clonidine
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Remifentanil+clonidine

INTERVENTIONS:
Drug: Remifentanil+clonidine — iv Remifentanil+ iv clonidine
  Other Names: Ultiva, Catapressan

SUMMARY:
The hypothesis is that systemic remifentanil and Clonidine act in a synergistic manner to relief acute main in an experimental human pain model. Of interest is also the effect of the combination on respiration, sedation and cognitive behavior.

DETAILED DESCRIPTION:
To examine the possible synergistic effects og systemic remifentanil and clonidine. Its effects on respiration, cognitive function and sedation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Relief of pain(VAS reduction) | Experimental

SECONDARY OUTCOMES:
Reduction in Minute ventilation | Experimental
Reduction in CO2 stimulated Minute Ventilation | experimental
Reduction in BIS score | Experimental
Performance on Stroop test | Experimental

CONTACTS AND LOCATIONS:
Overall Officials: Jon B Bergmann, Ass. Prof., Principal Investigator — Dep of Anesthesia and Intensive Care, Rikshospitalet-Radiumhospitalet Medical Center
Locations (1):
- Dep of Anesthesia and Intensive Care, Rikshospitalet-Radiumhospitalet Medical Center, Oslo, Norway